CLINICAL TRIAL: NCT06711185
Title: Effect of DAPAglifozin on MYOcardial Remodeling of Breast CANCER Patients Treated with Anthracycline Based Chemotherapy
Acronym: DAPA-MYOCANCER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Otavio Rizzi Coelho Filho, Professor (Assistant) at Unicamp, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 57488122.1.0000.5404
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Dapagliflozin; Anthracyclines; chemotherapy induced cardiomyopathy
MeSH Terms: conditions — Breast Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Standard chemotherapy treatment + Dapagliflozin 10mg/day.
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo Group (Placebo Comparator): Standard chemotherapy treatment + Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Patients in this group will receive 1 tablet of 10mg dapagliflozin daily for 9 months, starting 7-10 days before chemotherapy treatment.
  Arms: Dapagliflozin
Other: Placebo — Patients in this group will receive 1 placebo tablet per day, with identical characteristics to the group receiving dapagliflozin, for 9 months, starting 7-10 days before the start of chemotherapy treatment
  Arms: Placebo Group

SUMMARY:
Prospective, randomized, double-blind, controlled clinical trial to compare the effect of 9 months of treatment with dapagliflozin vs. placebo on anthracycline-induced cardiotoxicity in patients with breast cancer.

DETAILED DESCRIPTION:
Anthracycline-based chemotherapy is the standard treatment for several common cancer types, including breast cancer, lymphoma and sarcoma. However, within 12 months, up to 20% of the 1,000,000 patients worldwide treated with anthracyclines each year have a significant reduction in left ventricular ejection fraction (LVEF), leading to a three to six-fold higher rates of incident heart failure. Once established, anthracycline-induced heart failure carries a poor prognosis with a 2-year survival of only 40%.

Consistent data have established that sodium-glucose transport protein 2 (SGLT2) inhibitors reduce incident heart failure in patients without cancer. There is biological plausibility and animal data to support the hypothesis central to this proposal that SGLT2 will reduce anthracycline-induced cardiotoxicity (AIC). Anthracyclines increase inflammatory cytokines, increase cell death, increase myocardial fibrosis leading to a decrease in the LVEF. In animal and cellular models, SGLT2 inhibitors reduce inflammatory cytokines, increase cell viability, reduce myocardial fibrosis and prevent the decline in LVEF with anthracyclines. There are no preliminary clinical data testing whether SGLT2 inhibitors are cardioprotective during treatment with anthracyclines among patients with breast cancer.

We propose a single-center randomized double-blind placebo-controlled trial, in 80 patients, who will be randomized 1:1 to dapagliflozin 10mg/daily or placebo to determine whether dapagliflozin started prior to anthracyclines reduces AIC in patients breast cancer. The endpoint AIC will be defined as a 6% difference in the change in LVEF between groups within the first 9 months after the start of therapy. LVEF will be measured using the gold-standard, cardiac magnetic resonance (CMR), performed in an established core clinical trials laboratory by expert researchers.

Participants will be recruited over 2 years from a large volume academic oncology network. Myocardial fibrosis is a key intermediary that occurs prior to the development of LV dysfunction. CMR is the gold-standard imaging technique for fibrosis; therefore, to test whether the sub-acute development of myocardial fibrosis can predict the late occurrence of AIC and whether dapagliflozin reduces myocardial fibrosis, we also propose measuring the extent of fibrosis at baseline and 9 months.

We hypothesize that dapagliflozin will attenuate the anthracycline-induced increase in myocardial fibrosis. Secondary and exploratory outcomes will include significant changes in myocardial perfusion assessed by stress CMR, flow-mediated vasodilatation assessed by ultrasound, exercise capacity assessed by cardiopulmonary exercise test, and biomarkers.

If successful, this study will show that dapagliflozin started prior to anthracyclines will preserve the LVEF and will attenuate the anthracycline-induced cardiovascular toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 years old
* Breast cancer
* Chemotherapy as treatment planning and programmed cumulative dose equivalent to 240 mg/m2 of doxorubicin.

Exclusion Criteria:

* Contraindications for performing CMR exams, such as patients with pacemakers or cardiac defibrillators of any type, metal clips for cerebral aneurysms, cochlear implants, and ventriculoperitoneal bypass valves.
* Inability to perform CMR due to claustrophobia.
* Renal failure with a glomerular filtration rate < 30 ml/min/1.73 m2.
* Previous history of myocardial infarction, congestive heart failure, or myocardial revascularization, whether percutaneous or surgical.
* Previous history of significant valvular heart disease.
* Previous history of cardiomyopathies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female individuals (biological sex) with breast cancer.
Enrollment: 80 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricle ejection fraction | 36 weeks
  The primary outcome will be the 6% difference in the mean of left ventricle ejection fraction change, as assessed by CMR, between the placebo group and the dapagliflozin group

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Rizzi Coelho-Filho, MD, MPH, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Hospital de Clinicas da Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided